CLINICAL TRIAL: NCT04390230
Title: Inflatable Penile Prostheses : Predicting Factors of Pump Misuse and Unsatisfaction
Brief Title: Inflatable Penile Prostheses : Which Patients Can Correctly Use the Scrotal Pump ?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20Urobase01
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Surgery; Satisfaction; Penile Prosthesis; Complications
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with peniale implantation: All patients who underwent implantation with either Coloplast or Boston Scientific - AMS IPPs between 2014 and 2019, by 2 surgeons of the University Hospital of Nice, France.
  Interventions: Procedure: Penile prostheses implantation

INTERVENTIONS:
Procedure: Penile prostheses implantation — Penial implantation with either Coloplast or Boston Scientific - AMS IPPs between 2014 and 2019, by 2 surgeons of the University Hospital of Nice, France

SUMMARY:
Sexual health and satisfaction are well know as critical critera to assess quality of life, at any age. Among the multiple aspects of sexual health, erectile dysfunction (ED) is not anymore a fate, mainly thanks to the advent of phosphodiesterase type 5 (PDE5) inhibitors in 1998. Nevertheless, a significant part of patients are intolerant or does not respond to PDE5 inhibitors and thus are looking for other treatment options.

Since the first implantation of foreign material intracarvernosally in 1966 by Beheri, multiple modifications and enhancements were achieved in order to produce devices more reliable with a more natural appearance. First introduced in 1973 by Scott et al., inflatable prosthesis provides now high general satisfaction rates (69-94%), better than in malleable prostheses, except for few authors.

In addition to changes in materials and construction, the two main manufacturers of IPP, Boston scientific AMS (Marlborough, MA, USA) and Coloplast (Minneapolis, MN, USA), modernized the pump mechanism of their devices. Since the introduction of AMS IPP, three main pump formats have been used : the standard pump has been replaced in 2004 by the " Tactile " pump and then the " Momentary Squeeze " (MS) pump in 2006, smaller and easier to deflate by not requiring the patient to hold the deflation button throughout deflation. Coloplast also replaced in 2008 their " Genesis " pump by a " One Touch Release " (OTR) pump, and finally in 2014 by the current " Touch " pump, smaller, and presenting a biconcave deflation button, easier to find.

Despite all technological advances, appropriate pre-operative counselling and careful post-operative teachning, a significant part of patients has still difficulties to handle the pump and thus, does not use their IPP, regardless of any material malfunction. That situation obviously leads to patient's dissatisfaction and highlights the operating risks of a useless surgical procedure.

The purposes of this study were:to identify the risks factors, modifiable and non-modifiable, for patients' difficulty to inflate and/or deflate their device after IPP implantation, then to show a correlation between easy handling and post-operative satisfaction. And last but not least, to show an association between pre-operative pump pattern viewing and handling and post-operative easy handling. That information could help the physicians to improve the pre-operative selection of patients and to adapt the peri-operative care in order to improve patients satisfaction.

ELIGIBILITY:
All cases included were discussed and approved by a multidisciplinary team. Patients who underwent prosthesis replacement or second implantation were not included. We excluded patients who refused or were not able to answer our questionnaire, patients who provided unreliable answers, and patients that experimented a secondary malfunction of their IP.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent implantation with either Coloplast or Boston Scientific - AMS IPPs between 2014 and 2019, by 2 surgeons of the University Hospital of Nice, France.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-01-24 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
to identify the risks factors, modifiable and non-modifiable, for patients' difficulty to inflate and/or deflate their device after IPP implantation. | 3 months
  the statistical association between pump misusing, and a range of potentially relevant factors such as ages, BMI, model pump, inappropriate positionning or post operative complications

SECONDARY OUTCOMES:
to show a correlation between easy handling and post-operative satisfaction | 3 months
  statistical correlation between easy handling and post-operative satisfaction
to show an association between pre-operative pump pattern viewing and handling and post-operative easy handling | 3 months
  statistical association between pre-operative pump pattern viewing and handling and post-operative easy handling.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
No data sharing plan has been established.